CLINICAL TRIAL: NCT05190224
Title: Changes in Plantar Pressures and Ankle Range of Motion After the Technique of Neuromeningeal Mobilization of the Posterior Tibial Nerve, Deep Peroneal Nerve, Medial and Lateral Dorsocutaneous Nerve
Brief Title: Changes in Plantar Preassures and Ankle Range of Motion After the Technique of Neuromeningeal Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, Mayuben Private Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3010201915819
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Postural Balance; Rehabilitation; Foot; Therapy
Keywords: Platform; neural movilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental- (Experimental): All participants will be included in this arm
  Interventions: Other: Neural mobilization of the deep peroneal, posterior tibial and medial medial and lateral dorsocutaneous nerves.

INTERVENTIONS:
Other: Neural mobilization of the deep peroneal, posterior tibial and medial medial and lateral dorsocutaneous nerves. — In lateral decubitus the patient with the help of the clinician will perform neuromeningeal mobilization of the posterior tibial dorsocutaneous lateral, intermediate and medial nerves and deep peroneal nerve too.

SUMMARY:
Neuromeningeal mobilization or neurodynamics is a movement-based technique whose purpose is to restore peri- and intraneural homeostasis (1). It is based on principle that nerves have to lengthen and shorten to maintain normal muscle tension and range of motion (1) This technique has been shown to be effective in recovering tissue mobility (2), reducing pain in low back pain (3) and neck pain (1) and pain intensity in the elderly, and increasing joint range of motion and muscle flexibility (4 )

Regarding balance, sciatic nerve sliding has been shown to immediately improve balance to one leg ( dinamic balance) after application in a comparative study before and after (4,5)

No study has been realised in for the Posterior Tibial, Deep Peroneal, Medial Dorsocutaneous and Lateral Nerves, and no study has verificated standing balance and range of motion in ankle joint

DETAILED DESCRIPTION:
The study will consist of recording before and after applying the nerve mobilization exercise. Measurements will be made on the same day without the need to go at another time.

In this study, participants will be asked to stand on a pressure platform several times in a relaxed manner and with eyes open and closed before and after a neuromeningeal mobilization technique indicated for the treatment of pain in your feet. In addition, the mobility of the ankle will be measured with the knee flexed and stretched. The measurements or tests to be carried out are totally innocuous and do not carry any risk to your health and integrity.

Participants will have to remain barefoot for a maximum of 30 seconds, a total of 8 times on a pressure platform

ELIGIBILITY:
Inclusion criteria:

-Participants who arrived at the clinic presenting with pain in both heels and who were diagnosed with active or latent MTrP in bilateral flexor digitorum brevis, (2) these specific MTrPs were the only MTrPs diagnosed in limb or foot, (3) all participants had a normal body mass because obesity can affect plantar pressure distribution [28], and (4) and had an age range of 27.96 to 36.04 (95% confidence interval [CI]) because body mass could also affect plantar pressures.

Exclusion Criteria:

* (1) Diagnosis of lower limb injury, such as plantar fasciitis, tendinopathy, bursitis, ligament injuries [27], (2) a history of previous lower extremity surgery [28], (3) participants were required not to have undergone ankle stretching or any other treatment [23], (4) diabetes due to possible elevation of plantar pressure, [30], (5) deformities of the toes, such as hammer toes and hallux valgus due to their possible alteration in plantar pressure.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Variables of plantar pressures with platform before mobilization | Through study completion, an average of 2 days
  During 30 seconds we will record the plantar pressure variables in grams per square centimeter
Variable footprint plantar surface with platform before | Through study completion, an average of 2 days
  For 30 seconds we will record the area of the footprint in square centimeters.
Variables of plantar pressures with platform after mobilization | Through study completion, an average of 2 days
  During 30 seconds we will record the plantar pressure variables in grams per square centimeter
Variable footprint plantar surface with platform after mobilization | Through study completion, an average of 2 days
  For 30 seconds we will record the area of the footprint in square centimeters

CONTACTS AND LOCATIONS:
Overall Officials: EVA Martínez-Jimenez, Dr, Principal Investigator — Mayuben C
Locations (1):
- EVA MARIA Martínez, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
There will be no sharing plan